CLINICAL TRIAL: NCT00544934
Title: A Dose-ranging Study to Evaluate the Safety, Metabolism and Therapeutic Dosing of Three Multiple Dose Levels of GLY-230 in Healthy and Diabetic Subjects
Brief Title: Multiple Dose Trial of Anti-glycation Agent GLY-230 in Healthy and Diabetic Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Glycadia (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GLY-002
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — 2-(3-chlorophenylamino)phenylacetic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 250 mg (Experimental)
  Interventions: Drug: GLY-230
- 500 mg (Experimental)
  Interventions: Drug: GLY-230
- 750 mg (Experimental)
  Interventions: Drug: GLY-230
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GLY-230 — 125, 250 0r 375 mg bid for 14 days
  Arms: 250 mg; 500 mg; 750 mg
Other: Placebo — No drug administered
  Arms: Placebo

SUMMARY:
A dose-ranging study evaluating safety, metabolism and therapeutic dosing of three multiple dose levels of GLY-230 in healthy and diabetic subjects

ELIGIBILITY:
Inclusion Criteria:

* Nondiabetic and diabetic men age 18-55, engative drug screen, normal EKG, clinical chemistries. hematology parameters, HbA1c 7.5% if diabetic, give written informed consent

Exclusion Criteria:

* Sctive concomitant serious medical or surgical disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-02; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
glycated albumimin concentration | three weeks

SECONDARY OUTCOMES:
urine albumin | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Kennedy, M.D., Principal Investigator — University of Florida; Maria del Pilar Solano, M.D., Principal Investigator — University of Miami, Miami, Florida; Lis Cohen, D.O., Principal Investigator — Suncoast Clinical Research, New Port Richey, Florida